CLINICAL TRIAL: NCT05236166
Title: Rapid Versus Slow Withdrawal of Antiepileptic Monotherapy in 2-year Seizure-free Adult Patients With Epilepsy (RASLOW) Study: a Pragmatic Multicentre, Prospective, Randomized, Controlled Study
Brief Title: Multicentre Study on Rapid Versus Slow Withdrawal of Antiepileptic Monotherapy
Acronym: RASLOW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Magna Graecia (Other)
Collaborators: Ministry of Health, Italy (Other Government)
Responsible Party: Principal Investigator, Edoardo Ferlazzo, Professor, University Magna Graecia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GR-2013-02358677
Record Dates: First submitted 2022-01-18; First posted 2022-02-11 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-02

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — Anticonvulsants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rapid withdrawal (Other): Reduction by about 20 % of initial dosage every 15 days until complete discontinuation (total withdrawal time: 60 days).
  Interventions: Drug: Rapid withdrawal of antiepileptic
- Slow withdrawal (Other): Reduction by about 20 % of initial dosage every 40 days, until complete discontinuation (total withdrawal time: 160 days).
  Interventions: Drug: Slow withdrawal of antiepileptic

INTERVENTIONS:
Drug: Rapid withdrawal of antiepileptic — Reduction by about 20 % of initial dosage every 15 days until complete discontinuation (total withdrawal time: 60 days).
  Drugs: carbamazepine, lamotrigine, levetiracetam, oxcarbazepine, phenobarbital, phenytoin, topiramate, valproic acid, zonisamide
  Other Names: antiepileptic
  Arms: Rapid withdrawal
Drug: Slow withdrawal of antiepileptic — Slow withdrawal: reduction by about 20 % of initial dosage every 40 days, until complete discontinuation (total withdrawal time: 160 days).
  Drugs: carbamazepine, lamotrigine, levetiracetam, oxcarbazepine, phenobarbital, phenytoin, topiramate, valproic acid, zonisamide
  Other Names: antiepileptic
  Arms: Slow withdrawal

SUMMARY:
The main objective of the present study will be to establish whether a slow (within 160 days) or a rapid (within 60 days) withdrawal schedule of antiepileptic monotherapy influence relapse rate in adult patients with epilepsy, who have been seizure free for at least 2 years. Secondary objectives will be to establish the compliance rates with these two schedules and the differences in terms of severity of relapses, based on the occurrence of status epilepticus, seizure-related injuries and death.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of focal or generalized epilepsy (according to International League Against Epilepsy 1989 criteria)
* age at epilepsy onset of 16 years or older
* seizure freedom for at least 2 years
* treatment with one of the antiepilepsy drugs currently available for monotherapy in Italy: carbamazepine, lamotrigine, levetiracetam, oxcarbazepine, phenobarbital, phenytoin, topiramate, valproic acid zonisamide)
* adherence to the protocol and visit schedules.

Exclusion Criteria:

* inability to understand the aims or modalities of the study;
* current pregnancy or plans to become pregnant during withdrawal period;
* history of seizure relapse after discontinuation of treatment;
* history of psychogenic non-epileptic seizures (PNES);
* history of status epilepticus

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-04-26 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Time to seizure relapse | 365 days
  Time to recurrence of an epileptic seizure, assesed by telephone call and outpatients visits.

SECONDARY OUTCOMES:
Patients' compliance with the assigned withdrawal schedule | 365 days
  Compliance with the assigned withdrawal schedule (evaluated by telephone interview) and outpatients visits.
Severity of relapses and mortality | 365 days
  Severity of relapses, in terms of seizure-related injuries, status epilepticus (SE) during or after withdrawal period, and mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Regional Epilepsy Center, Presidio Riuniti, Magna Græcia University of Catanzaro, Reggio Calabria, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Del Felice A, Beghi E, Boero G, La Neve A, Bogliun G, De Palo A, Specchio LM. Early versus late remission in a cohort of patients with newly diagnosed epilepsy. Epilepsia. 2010 Jan;51(1):37-42. doi: 10.1111/j.1528-1167.2009.02141.x. Epub 2009 Jun 1. PMID 19490039
- [Background] Ranganathan LN, Ramaratnam S. Rapid versus slow withdrawal of antiepileptic drugs. Cochrane Database Syst Rev. 2006 Apr 19;(2):CD005003. doi: 10.1002/14651858.CD005003.pub2. PMID 16625621